CLINICAL TRIAL: NCT00274521
Title: A Randomized, Double-blind, Placebo Controlled 25-week Trial to Compare the Effect of Tiotropium Inhalation Capsuled (18 Mcg) Once Daily on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease (COPD) Participating in 8 Weeks of Pulmonary Rehabilitation.
Brief Title: Tiotropium (Spiriva) Rehabilitation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.230
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The study was designed to determine whether tiotropium inhalation capsules, compared to placebo, enhances the improvement in exercise tolerance seen in patients with chronic obstructive pulmonary disease (COPD) who participate in pulmonary rehabilitation. In addition, assessments of the effect of tiotropium on dyspnea and quality of life following pulmonary rehabilitation were taken.

ELIGIBILITY:
Inclusion Criteria:

History of COPD, FEV1 of less than or equal than 60% of predicted normal and less than or equal to 70% at Visit 1, Male or Female 40 years or greater, smoking history of more than 10 pack years (current or ex-smokers), patient can perform all study related tests, patients can inhale medication from HandiHaler and from meter dose inhaler, patients who would benefit from participation in a pulmonary rehab program and patients who had a medical clearance to participate in a pulmonary rehab program.

Exclusion Criteria:

Patients with significant diseases other than COPD, patients with clinically relevant abnormal baseline hematology, blood chemistry or urinalysis, all patients with SGOT greater than 80IU/L, bilirubin greater than 2.0 mg/dl or creatinine greater than 2.0 mg/dL, recent history of MI (6 months or less). any cardiac arrhythmia requiring drug therapy or has abeen hospitalized for heart failure with the past 3 years, active TB, history of CA or had treatment within the last 24 months, history of CF, bronchiectasis, interstitial lung disease or pulmonary thromboembolic disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2001-05; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in submaximal exercise tolerance (prior to treatment to after pulmonary rehabilitation) as measured by endurance time during a constant work rate treadmill exercise test at 80% of maximum work capacity | week 13

SECONDARY OUTCOMES:
Individual FEV1 measurement | week 4, 13, 25
Individual FVC measurement | week 4, 13, 25
St. George.s Hospital Respiratory Questionnaire (SGRQ) | week 4, 13, 25
Transition dyspnea index | week 4, 13, 25
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest) | week 4, 13, 25
Modified Borg scale | week 4, 13, 25
Amount of albuterol therapy used during the treatment period | 25 weeks
Number and length of exacerbations of COPD | 25 weeks
Physician's global evaluation | week 4, 13, 25
Patient peak flow rates twice daily | 25 weeks
Patient activity measurement | week 9, 13, 17, 21, 25
Change in submaximal exercise tolerance during constant work rate exercise | week 25
Change in submaximal exercise tolerance prior to and after pulmonary rehabilitation. | week 13
Occurrence of adverse events | 25 weeks
Pulse rate and blood pressure in conjunction with spirometry | 25 weeks
Changes in the physical examination from baseline and at the conclusion of patient participation in the trial | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Attention: John E. Hodgkin, M.D., Deer Park, California
  - Boehringer Ingelheim Investigational Site, Long Beach, California
  - UCLA School of Medicine, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - Harbor-UCLA Research and Education Institute, Torrance, California
  - Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Boehringer Ingelheim Investigational Site, Elk Grove Village, Illinois
  - UMass Memorial Medical Center, North Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durhan, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Everett, Washington